CLINICAL TRIAL: NCT06037525
Title: Clinical Evaluation of the PowerGlide™ Pro Midline Catheter
Acronym: Midline
Status: Completed | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: MIDLINE
Record Dates: First submitted 2023-06-01; First posted 2023-09-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pain; Catheter Infection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PowerGlide™ Pro Midline Catheter — Clinical evaluation of the PowerGlide™ Pro Midline Catheter in patients with vascular disease

SUMMARY:
Clinical evaluation of the PowerGlide™ Pro Midline Catheter in patients with vascular diseases

DETAILED DESCRIPTION:
Clinical evaluation of the PowerGlide™ Pro Midline Catheter in patients with vascular diseases. The selected patients are in need of a long-term i.v. therapy for reasons as antibiotic therapy or alprostadil therapy. The Midline catheter is a device, which is placed via Seldinger's technique to a vein usual on the upper extremity under ultrasound-control.

ELIGIBILITY:
Inclusion Criteria:

* need for i.v. therapy longer than 7 days
* poor peripheral vein status
* Administration of alprostadil

Exclusion Criteria:

* pending dialysis
* allergy to catheter material
* minor age
* life threatening conditions
* requirement for central venous catheter

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients in the vascular surgery department with above mentioned inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Dwelling Time | 0-29 days
  Length of catheter in situ time

SECONDARY OUTCOMES:
Administration of Alprostadil | 0-29 days
  Feasibility for the usage of Alprostadil measured by patients with development of thrombophlebitis or occlusion
Catheter Complications | 0-29 days
  Site complications as thrombophlebitis and occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hyhlik-Duerr, PhD, Study Director — University Hospital Augsburg Vascular Surgery
Locations (1):
- University Hospital Augsburg, Augsburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided